CLINICAL TRIAL: NCT03200730
Title: A Multicenter Randomized Controlled Trial of a Novel Family Dignity Intervention (FDI) for Asian Palliative Care
Brief Title: A Novel Family Dignity Intervention (FDI) for Asian Palliative Care
Acronym: FDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: HCA Hospice Care (Other); Dover Park Hospice Singapore (Unknown); National Cancer Centre, Singapore (Other); University of Manitoba (Other); University of Memphis (Other)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Assistant Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-2017-02-019
Record Dates: First submitted 2017-06-24; First posted 2017-06-27 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Palliative Care
Keywords: Family Dignity Intervention; Multicentre Randomized Control Trial; Palliative Care; End-of-Life Care

STUDY DESIGN:
Intervention Model Description: Randomization will be conducted by an independent statistician. Treatment allocation (Family-oriented Dignity Intervention or Control) will be performed by block randomization with a fixed block size of two; each block will comprise of two patients with comparable terminal illness, along with their family caregiver, to reduce potential confounding effects of different illness types. Allocation concealment is facilitated by using sequentially number opaque sealed envelopes for consecutive and eligible families. To reduce the risk of bias, the researcher opens the next envelope to ascertain which group the family has been allocated to after baseline measures have been collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Dignity Intervention group (Experimental): A standard framework of 12 FDI questions is given to patient-family dyads in the intervention group during baseline to provides them with the opportunity to think about their responses. During the intervention interview scheduled 2-3 days later, the FDI therapist follows that dyad's cues, help them to organize their thoughts, facilitate disclosure of cherished memories, and encourage the expression of appreciation. The interview is be recorded, quickly transcribed verbatim then edited into a coherent narrative. A second review session is arranged to review and finalize the edited transcript with the dyads. Once the "legacy" documents are ready, a final family sharing session is arranged for the dyads to share and read this document to each other and their loved ones.
  Interventions: Behavioral: Family Dignity Intervention group
- Control group (No Intervention): Patient-family dyads in the control group have at least four interviews with a designated member of the research team via psychosocial home visits. Completing the assessments and taking part in the interviews provides them with the opportunity to share their feelings and emotions along their illness trajectory. The extent to which they feel sharing is therapeutic is explored in the interview.

INTERVENTIONS:
Behavioral: Family Dignity Intervention group — A brief psychotherapeutic intervention offered to a family dyad (i.e., patient and one identified family caregiver) using narrative approach with life review elements. The purpose is to facilitate an open dialogue between the family dyad that strengthens family connectedness and emotional connection.
  Arms: Family Dignity Intervention group

SUMMARY:
Background: The lack of a holistic approach to palliative care can lead to a fractured sense of dignity at the end of life, resulting in depression, hopelessness, feelings of being a burden to others, and the loss of will to live among terminally-ill patients. Building on the clinical foundation of Dignity Therapy, together with the empirical understanding of dignity-related concerns of Asian families facing terminal-illness, a novel Family Dignity Intervention (FDI) has been developed for Asia palliative care. FDI comprises a recorded interview with a patient and his/her primary family caregiver, which is transcribed, edited into a legacy document, and return to the dyads for sharing with the rest of the patient's family. The aims of this study are to assess the feasibility, acceptability and potential effectiveness of FDI in reducing psychosocial, emotional, spiritual, and psychophysiological distress in community-dwelling and in-patient Asian older terminally-ill patients and their families living in Singapore.

Methods/Design: An open-label multicentre randomized controlled trial. 126 patient-family dyads are randomly allocated to one of two groups: (i) intervention group (FDI offered in addition to standard psychological care), and (ii) control group (standard psychological care). Both quantitative and qualitative outcomes are assessed in face-to-face interviews at baseline, three days and two week after intervention, and during an exit interview with family caregivers at two month post bereavement. Primary outcome measures include sense of dignity for patients and psychological distress for caregivers. Secondary outcomes include meaning in life, quality of life, spirituality, hopefulness, perceived support and psychophysiological well-being, as well as bereavement outcomes for caregivers. Qualitative data are analyzed using Framework method.

Discussion: To date, there is no available palliative care intervention for dignity enhancement in Asia. This first-of-its kind study develops and tests an evidence-based, family-driven psycho-socio-spiritual intervention for enhancing dignity and wellbeing among Asian patients and families facing mortality. It address a critical gap in the provision of holistic palliative care. The expected outcomes will contribute to advancements in both theories and practices of palliative care for Singapore and other Asian communities around the world.

DETAILED DESCRIPTION:
Study Design

This study adopts an open-label multicentre randomized controlled trial design comprising of two groups: (i) intervention group (Family Dignity Intervention offered in addition to standard psychological care), and (ii) control group (standard psychological care include emotional support and psychosocial home visits). Consenting participants including one patient and one family caregiver from one family unit (i.e. patient-family dyad) will be randomly allocated to one of these two groups after baseline assessment meetings have been conducted.

Study Sites

Study settings include two hospice service providers in Singapore. First, Dover Park Hospice (DPH) is a secular, nonprofit organization that offers both in-patient and homecare hospice services to terminally-ill patients and their families. It is one of the largest hospice service provider in the country with over 50 in-patient beds. Second, HCA Hospice Care (HCA) is a registered charity that offers daycare and homecare hospice services to terminally-ill patients and their families. With a head office and numerous satellite service stations across the country, it offers national wide services to all Singaporeans. Both DPH and HCA are funded publically and via donations, service admission are based on physician referrals and mean-testing mechanisms as ascribed by the Singapore Ministry of Health. Both service providers house a team of palliative care specialist including physicians, nurses, social workers and counselors to provide round-the-clock support to individuals and families facing the end of life.

Participants

The sample comprises 126 Asian families in Singapore. Each family includes a patient-family dyad: (i) one older terminally-ill patients, and (ii) one identified family member whom the patient considers to be his or her primary or trusted caregiver. Participants are recruited through the in-patient, daycare and homecare hospice service units of DPH and HCA.

Recruitment, assessment, intervention and follow-up procedures

Appointed research nurses of DPH and HCA are asked to distribute research information pamphlets to all patients and family caregivers eligible for the study, based on their clinical assessments of patients using the Karnofsky Performance Status Scale; patients who received a score of 20 or below are considered too ill and ineligible to participate. At least one week is given for full consideration to participate in the study, after which, the research nurses contact each eligible family to seek their verbal consent for study participation. Once verbal consent is obtained, a simple information sheet containing the names and contact details of the patient-family dyad are forwarded to a member of the research team. The responsible researcher then contacts the patient-family dyad via telephone to organize a convenient time for the first baseline assessment meeting.

The first meeting is attended by the appointed FDI therapist, as well as responsible researcher who will (i) explains the study to the patient-family dyad; (ii) answer any questions they may have about their participation; (iii) checks that they have fully understood the implications of the study before obtaining written consent. As a final check, the researcher screens patients with the Mini-Mental State Exam to assess cognitive functioning, and those who scored below 18 are considered unfit to participate. In such cases patient-family dyads are excluded. This will be done sensitively, whereby the researcher and the FDI therapist spend some time chatting with the patient-family dyads about neutral topics before ending the meeting. This approach has worked successfully in previous studies of similar nature.

For patient-family dyads who are deemed fit to participate after the final check, the researcher conducts a baseline assessment with patients and caregivers individually, then open the next envelop in sequence to ascertain group allocation. Dyads assigned to the control group are reminded that they will receive three to four psychosocial visits from the research team, through which they will have the opportunity to share their feelings along their illness trajectory as well as their views on taking part in the study. Dyads assigned to the intervention group are given two sets of FDI framework questions, one for patients and one for caregivers, so that they have an opportunity to think and discuss about their responses. After a brief framing session conducted by the FDI therapist, a time will be arrange for the intervention interview within the next two to three days.

After the intervention interview is completed, the recorded transcript has been edited and finalized by the patient-family dyad, the FDI therapist sets up a time for a family sharing session in which the 'legacy' document is shared with selected members of the patients' family. A hard copy of the legacy document is also be given the patient-family dyad for safekeeping.

ELIGIBILITY:
Inclusion Criteria:

* Terminally-ill patients with a life expectancy of no more than 6 months
* Living in the community and receiving hospice home-and-day care services, OR, residing in long-term-care or hospice facilities and receiving hospice palliative care
* Score 30 and above on Karnofsky Performance Status Scale
* Score 18 and above on Mini-Mental State Examination (MMSE)
* Able to speak English, Mandarin, or Cantonese

Exclusion Criteria:

* Too ill to participate
* Unable to provide informed consent either due to cognitive problems or severity of illness
* Perform poorly on Karnofsky Performance Status Scale (i.e., scoring less than 30)
* Perform poorly on MMSE (i.e., scoring less than 18)
* Having moderate or severe cognitive impairment
* Unable to understand English, Mandarin, or Cantonese

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline 'Patient Dignity Inventory (PDI)' at 14 days [T2] and 4 weeks [T3] follow-up. | For patients, it will be assessed at baseline [T1], 14 days [T2] and four weeks [T3] follow-up.
  This 25-item measure evolved directly from the dignity model and comprised of questions relevant to the physical, psychosocial, existential and spiritual domain of end-of-life concern or distress.
Change from Baseline 'Patient Health Questionnaire' at 14 days [T2] and 4 week [T3] follow-up, and 2 months [T4] post bereavement. | For Caregivers, it will be assessed at baseline [T1], 14 days [T2] and four weeks [T3] follow-up, as well as two months [T4] following bereavement.
  This 9-item questionnaire measures patients' psychological distress.

SECONDARY OUTCOMES:
Change from Baseline 'Patient Health Questionnaire' at T2 and T3. | For patients, this will be assessed at baseline [T1], 14 days [T2] and four weeks [T3] follow-up.
  This 9-item questionnaire measures patients' psychological distress.
Change from Baseline 'Caregiver Self-Assessment' at T2, T3 and T4. | For Caregivers, this will be assessed at baseline [T1], two weeks [T2] and eight weeks [T3] follow-up, as well as two months [T4] following bereavement.
  This 18-item questionnaire measures family caregivers' well-being.
Change from Baseline 'Cancer Coherence Scale' at T2, T3 and T4. | For Patients, this will be assessed at baseline [T1], 14 days [T2] and four weeks [T3] follow-up. For Caregivers, this will be assessed at baseline [T1], two weeks [T2] and four weeks [T3] follow-up, as well as two months [T4] following bereavement.
  This 11-item questionnaire measures patients' and family caregivers' perceived meaning in life.
Change from Baseline 'World Health Organization Quality of Life Scale-8' at T2, T3 and T4. | For Patients, this will be assessed at baseline [T1], 14 days [T2] and four weeks [T3] follow-up. For Caregivers, this will be assessed at baseline [T1], two weeks [T2] and four weeks [T3] follow-up, as well as two months [T4] following bereavement.
  This 11-item questionnaire measures patients' and family caregivers' perceived quality of life.
Change from Baseline 'FACIT Spiritual Well-being Scale' at T2, T3 and T4. | For Patients, this will be assessed at baseline [T1], 14 days [T2] and four weeks [T3] follow-up. For Caregivers, this will be assessed at baseline [T1], two weeks [T2] and four weeks [T3] follow-up, as well as two months [T4] following bereavement.
  This 12-item questionnaire measures patients' and family caregivers' spirituality.
Change from Baseline 'Herth Hope Index' at T2, T3 and T4. | For Patients, this will be assessed at baseline [T1], 14 days [T2] and four weeks [T3] follow-up. For Caregivers, this will be assessed at baseline [T1], two weeks [T2] and four weeks [T3] follow-up, as well as two months [T4] following bereavement.
  This 12-item questionnaire measures patients' and family caregivers' hopefulness.
Change from Baseline 'Inventory of Social Support' at T2 and T3, as well as T4 for caregivers only. | For Patients, this will be assessed at baseline [T1], 14 days [T2] and four weeks [T3] follow-up. For Caregivers, this will be assessed at baseline [T1], two weeks [T2] and four weeks [T3] follow-up, as well as two months [T4] following bereavement.
  This 5-item questionnaire measures patients' and family caregivers' perceived social support.
Brief Grief Questionnaire | This will serve as a secondary outcome for family caregivers only, This will be assessed two months [T4] following family caregivers' bereavement.
  This 5-item questionnaire measures family caregivers' experience with grief.
Core Bereavement Items | This will serve as a secondary outcome for family caregivers only, This will be assessed two months [T4] following family caregivers' bereavement.
  This 17-item questionnaire measures family caregivers' experience with bereavement.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Ho, PhD, EdD, Principal Investigator — Nanyang Technological University
Locations (2):
- Singapore (2):
  - Dover Park Hospice Care, Singapore
  - HCA Hospice Care, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho AH, Chan CL, Leung PP, Chochinov HM, Neimeyer RA, Pang SM, Tse DM. Living and dying with dignity in Chinese society: perspectives of older palliative care patients in Hong Kong. Age Ageing. 2013 Jul;42(4):455-61. doi: 10.1093/ageing/aft003. Epub 2013 Feb 25. PMID 23443510
- [Background] Ho AH, Leung PP, Tse DM, Pang SM, Chochinov HM, Neimeyer RA, Chan CL. Dignity amidst liminality: healing within suffering among Chinese terminal cancer patients. Death Stud. 2013 Nov-Dec;37(10):953-70. doi: 10.1080/07481187.2012.703078. PMID 24517523
- [Background] Chochinov HM, Hack T, Hassard T, Kristjanson LJ, McClement S, Harlos M. Dignity therapy: a novel psychotherapeutic intervention for patients near the end of life. J Clin Oncol. 2005 Aug 20;23(24):5520-5. doi: 10.1200/JCO.2005.08.391. PMID 16110012
- [Background] Chochinov HM, Hack T, McClement S, Kristjanson L, Harlos M. Dignity in the terminally ill: a developing empirical model. Soc Sci Med. 2002 Feb;54(3):433-43. doi: 10.1016/s0277-9536(01)00084-3. PMID 11824919
- [Derived] Ho AHY, Car J, Ho MR, Tan-Ho G, Choo PY, Patinadan PV, Chong PH, Ong WY, Fan G, Tan YP, Neimeyer RA, Chochinov HM. A novel Family Dignity Intervention (FDI) for enhancing and informing holistic palliative care in Asia: study protocol for a randomized controlled trial. Trials. 2017 Dec 4;18(1):587. doi: 10.1186/s13063-017-2325-5. PMID 29202863